CLINICAL TRIAL: NCT02214303
Title: The Role of Th9 Cells Expression and Eosinophils Activity in the Course of Allergic Airway Diseases
Brief Title: The Role of Th9 Cells and Eosinophils Activity in Allergic Airway Diseases
Acronym: SAIRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Raimundas Sakalauskas, prof., dr., Lithuanian University of Health Sciences
Other Study IDs: SAIRA-1017/2012
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Allergic Asthma; Allergic Rhinitis
Keywords: Allergic asthma; Allergic rhinitis; Healthy subjects
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum and peripheral blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Allergic asthma: Allergic asthma (sensibilisation to D. pteronyssinus, 5 grass mixture allergens or birch pollen allergens)
- Allergic rhinitis: allergic rhinitis patients (sensibilisation to D. pteronyssinus, 5 grass mixture allergens or birch pollen allergens)
- Control group: Healthy subjects

SUMMARY:
The prevalence of allergic diseases, especially airway allergic diseases, has increased dramatically over the last twenty years all over the world including Lithuania. Allergic diseases are associated with significantly reduced quality of life and can sometimes cause death. Allergic diseases have turned into an important economic and social burden and nowadays take a more and more important place in the health system. Despite all intensive investigations, the pathogenesis of allergic airway diseases still remains unclear. As allergic diseases have a systemic pattern and multicomponent pathogenesis, it is important to investigate not individual cells, but examine various inflammatory cells instead, including their biological products and possible cellular interactions along the course of allergic diseases. This research focuses on the cells that are claimed to be important in the pathogenesis of allergic airway diseases, i.e. a newly found effector T helper cell subset (Th9 cells), which still lacks deeper investigation, and the main inflammatory cell, eosinophil. This study aims at determining the importance the way the Th9 lymphocytes perform, the eosinophil's activity, as well as molecular factors affecting these cells has in the process of prognostication of allergic airway diseases, namely allergic rhinitis and allergic asthma. An allergen challenge test will be performed in order to define the meaning of pathogenetic changes. The results of this research may reveal useful information in the course of allergic diseases and may be valuable when creating strategic principles of prophylaxis. The findings could be used for prevention and early diagnostics of allergic diseases and it could also open doors to discovering new and effective treatment.

ELIGIBILITY:
I. Inclusion criteria:

1. Men and women between the ages of 18-50 years;
2. Allergic asthma (skin prick test positive for D. pteronyssinus, 5 grass mixture or birch pollen);
3. Symptoms more than one year;
4. Positive Bronchial challenge with methacholine or documented completely reversible bronchial obstruction;
5. Stable lung function (FEV1≥70 perc.);
6. Allergic rhinitis diagnosed according ARIA criteria.
7. Postmenopausal women. Premenopausal women if pregnancy test is negative
8. Healthy (subjects who are not sick with acute or chronic inflammatory, infectious, oncologic or immune diseases) - control group
9. Participants who gave his/her informed written consent.

II. Exclusion criteria

1. Asthma and rhinitis exacerbation;
2. Clinically significant permanent allergy symptoms (ex. cat or dog dander induced allergy);
3. Active airway infection 1 month prior the study;
4. Used medicaments:

   1. Inhaled glucocorticoids intake 1 month prior the study;
   2. Antihistamines intake 7 days prior the study;
   3. Short acting β2 agonists 12 hours prior the study;
   4. Long acting β2 agonists 2 days prior the study;
   5. Leukotriene receptor antagonists prior 14 days;
5. If the histamine mean wheal diameter is <= 3 mm or control mean wheal diameter is >= 3 mm;
6. Psychiatric disorders;
7. Alcohol or narcotic abuse;
8. Pregnancy.
9. Breast-feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Allergic asthma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Th9 cells and eosinophil apoptosis | 24 hours after bronchial allergen challenge
  Blood and sputum eosinophils also peripheral blood th9 cells will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Raimundas Sakalauskas, Prof., dr., Study Chair — Lithuanian University of Health Sciences, Pulmonology and Immunology department
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Derived] Hoppenot D, Malakauskas K, Lavinskiene S, Sakalauskas R. p-STAT6, PU.1, and NF-kappaB are involved in allergen-induced late-phase airway inflammation in asthma patients. BMC Pulm Med. 2015 Oct 14;15:122. doi: 10.1186/s12890-015-0119-7. PMID 26466682